CLINICAL TRIAL: NCT04242966
Title: The Effect of Higher Protein Dosing in Critically Ill Patients: A Multicenter Registry-based Randomized Trial: The EFFORT Ultrasound a Sub-study
Brief Title: The Effect of Higher Protein Dosing in Critically Ill Patients Ultrasound a Sub-study
Acronym: EFFORTUS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never started. Operational issues prevented study from rolling out
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: The EFFORT Ultrasound
Record Dates: First submitted 2019-05-24; First posted 2020-01-27 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Critical Illness; Malnutrition
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive a usual protein/amino acid dose (≤1.2 g/kg/d)
  Interventions: Other: Usual Care; Other: Ultrasound measure
- Higher Protein/Amino Acid Group (Active Comparator): Patients will receive a higher protein/amino acid dose (≥2.2 g/kg/d).
  Interventions: Other: Higher Protein/Amino Acid Group; Other: Ultrasound measure

INTERVENTIONS:
Other: Usual Care — Protein targets will be set using pre-ICU dry actual weight. For patients with BMI >30, ideal body weight based on a BMI of 25 will be used. We will endorse the guidelines for energy targets set forth by ASPEN/SCCM, especially as it pertains to the obese patient.
  Arms: Usual Care
Other: Higher Protein/Amino Acid Group — Protein targets will be set using pre-ICU dry actual weight. For patients with BMI >30, ideal body weight based on a BMI of 25 will be used. We will endorse the guidelines for energy targets set forth by ASPEN/SCCM, especially as it pertains to the obese patient.
  Arms: Higher Protein/Amino Acid Group
Other: Ultrasound measure — Patients will undergo the ultrasound measures at baseline (within 24 hours of randomization, day 10 days post randomization (if still in hospital) and just prior to hospital discharge. In the event that hospital discharge is prior to day 10, the day 10 measure will not be done.

SUMMARY:
The investigators will evaluate the effects of of higher protein/amino acid dosing (≥2.2 g/kg/d) vs usual care of protein/amino acid dosing (≤1.2 g/kg/d) over muscle mass in nutritionally high risk ill patients.

DETAILED DESCRIPTION:
The EFFORT Ultrasound (US) is a sub study of the parent EFFORT trial; a multi-center, pragmatic, volunteer-driven, registry-based, randomized, clinical trial of 4000 nutritionally high-risk critically ill patients in the intensive care unit. Patients will be randomized to 1 of 2 treatment groups: a usual care prescription (≤1.2 g/kg/d) or a higher prescription (≥2.2 g/kg/d) of protein. Other than the protein amount the patient is randomized to, the remainder of care provided to randomized patient will be at the discretion of ICU providers.

In both groups, targets will be achieved through any combination of enteral nutrition (high protein content in high group if available), protein supplements, and parenteral nutrition or amino acids only (as clinically available). The only difference between the 2 groups is the protein targets that are set. Similar efforts should be used in both groups to achieve at least 80% of these targets. The remainder of care provided to eligible patients will be at the discretion of ICU providers.

Patients in the US sub-study will undergo the US measures at baseline (within 24 hours of randomization, 10 days post randomization (if still in hospital) and just prior to hospital discharge. In the event that hospital discharge is prior to day 10, the day 10 measure will not be done. To ensure standardization and quality in the measures, we have created high quality training materials and will have US films sent centrally to abstract all measurements. In the first 10 patients enrolled in the US sub-study, participating sites will conduct a run-in phase where their submitted data will be evaluated for quality and reliability (both intra and inter-rater reliability) to ensure subsequent measures are of high quality. Nutritional and clinical data for these patients will be included in the parent EFFORT trial but the US measures may be omitted if quality is poor.

The investigator has posed the following research question:

Primary Sub Study Research Question:

In critically ill patients with nutrition 'risk factors', what is the effect of prescribing a higher dose (≥2.2 grams/kg/day) of protein/amino acid administration compared to the usual care prescription (≤1.2 gram/kg/day) on muscle mass and quality, and 60 day mortality?

The proposed hypothesis:

Compared to receiving the usual care of protein/amino acids, the administration of a higher dose of protein/amino acids (a consequence of having a higher prescription) to nutritionally high-risk critically ill patients will be associated with greater muscle mass, improved survival and a quicker rate of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. - ≥18 years old
2. - Nutritionally 'high-risk' (meeting one of the below criteria)

   1. Low (≤25) or High BMI (≥35)
   2. Moderate to severe malnutrition (as defined by local assessments). We will document the means by which sites are making this determination and capture the elements of the assessment (history of weight loss, history of reduced oral intake, etc.).
   3. Frailty (Clinical Frailty Scale 5 or more from proxy)
   4. Sarcopenia- (SARC-F score of 4 or more from proxy)
   5. From point of screening, projected duration of mechanical ventilation >4 days
3. - Requiring mechanical ventilation with actual or expected total duration of mechanical ventilation >48 hours

Exclusion Criteria:

1. >96 continuous hours of mechanical ventilation before screening
2. Expected death or withdrawal of life-sustaining treatments within 7 days from screening
3. Pregnant
4. The responsible clinician feels that the patient either needs low or high protein
5. Patient requires parenteral nutrition only and site does not have products to reach the high protein dose group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of Muscle mass of the quadriceps from baseline to day 10 post randomization | at baseline (within 24 hours of randomization, day 10 days post randomization (if still in hospital) and just prior to hospital discharge. In the event that hospital discharge is prior to day 10, the day 10 measure will not be done
  Using ultrasound of quadriceps
Change of Muscle quality of the quadriceps from baseline to day 10 post randomization | at baseline (within 24 hours of randomization, day 10 days post randomization (if still in hospital) and just prior to hospital discharge. In the event that hospital discharge is prior to day 10, the day 10 measure will not be done
  Using ultrasound of quadriceps

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoffer LJ, Bistrian BR. Appropriate protein provision in critical illness: a systematic and narrative review. Am J Clin Nutr. 2012 Sep;96(3):591-600. doi: 10.3945/ajcn.111.032078. Epub 2012 Jul 18. PMID 22811443
- [Background] Heyland DK, Cahill N, Day AG. Optimal amount of calories for critically ill patients: depends on how you slice the cake! Crit Care Med. 2011 Dec;39(12):2619-26. doi: 10.1097/CCM.0b013e318226641d. PMID 21705881
- [Background] Heyland DK, Weijs PJ, Coss-Bu JA, Taylor B, Kristof AS, O'Keefe GE, Martindale RG. Protein Delivery in the Intensive Care Unit: Optimal or Suboptimal? Nutr Clin Pract. 2017 Apr;32(1_suppl):58S-71S. doi: 10.1177/0884533617691245. Epub 2017 Mar 1. PMID 28388372
- [Background] James S, Rao SV, Granger CB. Registry-based randomized clinical trials--a new clinical trial paradigm. Nat Rev Cardiol. 2015 May;12(5):312-6. doi: 10.1038/nrcardio.2015.33. Epub 2015 Mar 17. PMID 25781411
- [Background] Frobert O, Lagerqvist B, Olivecrona GK, Omerovic E, Gudnason T, Maeng M, Aasa M, Angeras O, Calais F, Danielewicz M, Erlinge D, Hellsten L, Jensen U, Johansson AC, Karegren A, Nilsson J, Robertson L, Sandhall L, Sjogren I, Ostlund O, Harnek J, James SK; TASTE Trial. Thrombus aspiration during ST-segment elevation myocardial infarction. N Engl J Med. 2013 Oct 24;369(17):1587-97. doi: 10.1056/NEJMoa1308789. Epub 2013 Aug 31. PMID 23991656
- [Background] Jolly SS, Cairns JA, Yusuf S, Meeks B, Pogue J, Rokoss MJ, Kedev S, Thabane L, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Steg PG, Bernat I, Xu Y, Cantor WJ, Overgaard CB, Naber CK, Cheema AN, Welsh RC, Bertrand OF, Avezum A, Bhindi R, Pancholy S, Rao SV, Natarajan MK, ten Berg JM, Shestakovska O, Gao P, Widimsky P, Dzavik V; TOTAL Investigators. Randomized trial of primary PCI with or without routine manual thrombectomy. N Engl J Med. 2015 Apr 9;372(15):1389-98. doi: 10.1056/NEJMoa1415098. Epub 2015 Mar 16. PMID 25853743
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Background] Nicolo M, Heyland DK, Chittams J, Sammarco T, Compher C. Clinical Outcomes Related to Protein Delivery in a Critically Ill Population: A Multicenter, Multinational Observation Study. JPEN J Parenter Enteral Nutr. 2016 Jan;40(1):45-51. doi: 10.1177/0148607115583675. Epub 2015 Apr 21. PMID 25900319
- [Background] Alberda C, Gramlich L, Jones N, Jeejeebhoy K, Day AG, Dhaliwal R, Heyland DK. The relationship between nutritional intake and clinical outcomes in critically ill patients: results of an international multicenter observational study. Intensive Care Med. 2009 Oct;35(10):1728-37. doi: 10.1007/s00134-009-1567-4. Epub 2009 Jul 2. PMID 19572118
- [Background] Heyland DK, Stephens KE, Day AG, McClave SA. The success of enteral nutrition and ICU-acquired infections: a multicenter observational study. Clin Nutr. 2011 Apr;30(2):148-55. doi: 10.1016/j.clnu.2010.09.011. Epub 2010 Oct 25. PMID 20971534
- [Background] Liebau F, Sundstrom M, van Loon LJ, Wernerman J, Rooyackers O. Short-term amino acid infusion improves protein balance in critically ill patients. Crit Care. 2015 Mar 12;19(1):106. doi: 10.1186/s13054-015-0844-6. PMID 25882298
- [Background] Hsieh LC, Chien SL, Huang MS, Tseng HF, Chang CK. Anti-inflammatory and anticatabolic effects of short-term beta-hydroxy-beta-methylbutyrate supplementation on chronic obstructive pulmonary disease patients in intensive care unit. Asia Pac J Clin Nutr. 2006;15(4):544-50. PMID 17077073
- [Background] Wei X, Day AG, Ouellette-Kuntz H, Heyland DK. The Association Between Nutritional Adequacy and Long-Term Outcomes in Critically Ill Patients Requiring Prolonged Mechanical Ventilation: A Multicenter Cohort Study. Crit Care Med. 2015 Aug;43(8):1569-79. doi: 10.1097/CCM.0000000000001000. PMID 25855901
- [Background] Allingstrup MJ, Esmailzadeh N, Wilkens Knudsen A, Espersen K, Hartvig Jensen T, Wiis J, Perner A, Kondrup J. Provision of protein and energy in relation to measured requirements in intensive care patients. Clin Nutr. 2012 Aug;31(4):462-8. doi: 10.1016/j.clnu.2011.12.006. Epub 2011 Dec 29. PMID 22209678
- [Background] Weijs PJ, Looijaard WG, Beishuizen A, Girbes AR, Oudemans-van Straaten HM. Early high protein intake is associated with low mortality and energy overfeeding with high mortality in non-septic mechanically ventilated critically ill patients. Crit Care. 2014 Dec 14;18(6):701. doi: 10.1186/s13054-014-0701-z. PMID 25499096
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Casaer MP, Wilmer A, Hermans G, Wouters PJ, Mesotten D, Van den Berghe G. Role of disease and macronutrient dose in the randomized controlled EPaNIC trial: a post hoc analysis. Am J Respir Crit Care Med. 2013 Feb 1;187(3):247-55. doi: 10.1164/rccm.201206-0999OC. Epub 2012 Nov 29. PMID 23204255
- [Background] Schetz M, Casaer MP, Van den Berghe G. Does artificial nutrition improve outcome of critical illness? Crit Care. 2013 Feb 1;17(1):302. doi: 10.1186/cc11828. PMID 23375069
- [Background] Casaer MP, Van den Berghe G. Nutrition in the acute phase of critical illness. N Engl J Med. 2014 Mar 27;370(13):1227-36. doi: 10.1056/NEJMra1304623. No abstract available. PMID 24670169
- [Background] Braunschweig CL, Freels S, Sheean PM, Peterson SJ, Perez SG, McKeever L, Lateef O, Gurka D, Fantuzzi G. Role of timing and dose of energy received in patients with acute lung injury on mortality in the Intensive Nutrition in Acute Lung Injury Trial (INTACT): a post hoc analysis. Am J Clin Nutr. 2017 Feb;105(2):411-416. doi: 10.3945/ajcn.116.140764. Epub 2016 Dec 14. PMID 27974311
- [Background] Arabi YM, Aldawood AS, Haddad SH, Al-Dorzi HM, Tamim HM, Jones G, Mehta S, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Afesh L; PermiT Trial Group. Permissive Underfeeding or Standard Enteral Feeding in Critically Ill Adults. N Engl J Med. 2015 Jun 18;372(25):2398-408. doi: 10.1056/NEJMoa1502826. Epub 2015 May 20. Erratum In: N Engl J Med. 2015 Sep 24;373(13):1281. doi: 10.1056/NEJMx150028. PMID 25992505
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Background] Needham DM, Dinglas VD, Bienvenu OJ, Colantuoni E, Wozniak AW, Rice TW, Hopkins RO; NIH NHLBI ARDS Network. One year outcomes in patients with acute lung injury randomised to initial trophic or full enteral feeding: prospective follow-up of EDEN randomised trial. BMJ. 2013 Mar 19;346:f1532. doi: 10.1136/bmj.f1532. PMID 23512759
- [Background] Doig GS, Simpson F, Sweetman EA, Finfer SR, Cooper DJ, Heighes PT, Davies AR, O'Leary M, Solano T, Peake S; Early PN Investigators of the ANZICS Clinical Trials Group. Early parenteral nutrition in critically ill patients with short-term relative contraindications to early enteral nutrition: a randomized controlled trial. JAMA. 2013 May 22;309(20):2130-8. doi: 10.1001/jama.2013.5124. PMID 23689848
- [Background] Doig GS, Simpson F, Bellomo R, Heighes PT, Sweetman EA, Chesher D, Pollock C, Davies A, Botha J, Harrigan P, Reade MC. Intravenous amino acid therapy for kidney function in critically ill patients: a randomized controlled trial. Intensive Care Med. 2015 Jul;41(7):1197-208. doi: 10.1007/s00134-015-3827-9. Epub 2015 Apr 30. PMID 25925203
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Jie B, Jiang ZM, Nolan MT, Zhu SN, Yu K, Kondrup J. Impact of preoperative nutritional support on clinical outcome in abdominal surgical patients at nutritional risk. Nutrition. 2012 Oct;28(10):1022-7. doi: 10.1016/j.nut.2012.01.017. Epub 2012 Jun 5. PMID 22673593
- [Background] Heyland DK, Dhaliwal R, Jiang X, Day AG. Identifying critically ill patients who benefit the most from nutrition therapy: the development and initial validation of a novel risk assessment tool. Crit Care. 2011;15(6):R268. doi: 10.1186/cc10546. Epub 2011 Nov 15. PMID 22085763
- [Background] Rahman A, Hasan RM, Agarwala R, Martin C, Day AG, Heyland DK. Identifying critically-ill patients who will benefit most from nutritional therapy: Further validation of the "modified NUTRIC" nutritional risk assessment tool. Clin Nutr. 2016 Feb;35(1):158-162. doi: 10.1016/j.clnu.2015.01.015. Epub 2015 Jan 28. PMID 25698099
- [Background] Compher C, Chittams J, Sammarco T, Nicolo M, Heyland DK. Greater Protein and Energy Intake May Be Associated With Improved Mortality in Higher Risk Critically Ill Patients: A Multicenter, Multinational Observational Study. Crit Care Med. 2017 Feb;45(2):156-163. doi: 10.1097/CCM.0000000000002083. PMID 28098623
- [Background] Mukhopadhyay A, Henry J, Ong V, Leong CS, Teh AL, van Dam RM, Kowitlawakul Y. Association of modified NUTRIC score with 28-day mortality in critically ill patients. Clin Nutr. 2017 Aug;36(4):1143-1148. doi: 10.1016/j.clnu.2016.08.004. Epub 2016 Aug 12. PMID 27582120
- [Background] Mendes R, Policarpo S, Fortuna P, Alves M, Virella D, Heyland DK; Portuguese NUTRIC Study Group. Nutritional risk assessment and cultural validation of the modified NUTRIC score in critically ill patients-A multicenter prospective cohort study. J Crit Care. 2017 Feb;37:45-49. doi: 10.1016/j.jcrc.2016.08.001. Epub 2016 Aug 10. PMID 27621112
- [Background] Rosa M, Heyland DK, Fernandes D, Rabito EI, Oliveira ML, Marcadenti A. Translation and adaptation of the NUTRIC Score to identify critically ill patients who benefit the most from nutrition therapy. Clin Nutr ESPEN. 2016 Aug;14:31-36. doi: 10.1016/j.clnesp.2016.04.030. Epub 2016 May 21. PMID 28531396
- [Background] Arabi YM, Aldawood AS, Al-Dorzi HM, Tamim HM, Haddad SH, Jones G, McIntyre L, Solaiman O, Sakkijha MH, Sadat M, Mundekkadan S, Kumar A, Bagshaw SM, Mehta S; PermiT trial group. Permissive Underfeeding or Standard Enteral Feeding in High- and Low-Nutritional-Risk Critically Ill Adults. Post Hoc Analysis of the PermiT Trial. Am J Respir Crit Care Med. 2017 Mar 1;195(5):652-662. doi: 10.1164/rccm.201605-1012OC. PMID 27589411
- [Background] Connolly B, MacBean V, Crowley C, Lunt A, Moxham J, Rafferty GF, Hart N. Ultrasound for the assessment of peripheral skeletal muscle architecture in critical illness: a systematic review. Crit Care Med. 2015 Apr;43(4):897-905. doi: 10.1097/CCM.0000000000000821. PMID 25559437
- [Background] Tillquist M, Kutsogiannis DJ, Wischmeyer PE, Kummerlen C, Leung R, Stollery D, Karvellas CJ, Preiser JC, Bird N, Kozar R, Heyland DK. Bedside ultrasound is a practical and reliable measurement tool for assessing quadriceps muscle layer thickness. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):886-90. doi: 10.1177/0148607113501327. Epub 2013 Aug 26. PMID 23980134
- [Background] Paris MT, Mourtzakis M, Day A, Leung R, Watharkar S, Kozar R, Earthman C, Kuchnia A, Dhaliwal R, Moisey L, Compher C, Martin N, Nicolo M, White T, Roosevelt H, Peterson S, Heyland DK. Validation of Bedside Ultrasound of Muscle Layer Thickness of the Quadriceps in the Critically Ill Patient (VALIDUM Study). JPEN J Parenter Enteral Nutr. 2017 Feb;41(2):171-180. doi: 10.1177/0148607116637852. Epub 2016 Jul 11. PMID 26962061
- [Background] Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, Annoni R, Puthucheary Z, Gordon IR, Morris PE, Denehy L. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care. 2015 Oct;30(5):1151.e9-14. doi: 10.1016/j.jcrc.2015.05.024. Epub 2015 Jun 3. PMID 26211979
- [Background] See www.criticalcarenutrition.com for most recent version of the Canadian Critical Care Nutrition Guidelines
- [Background] Martin CM, Doig GS, Heyland DK, Morrison T, Sibbald WJ; Southwestern Ontario Critical Care Research Network. Multicentre, cluster-randomized clinical trial of algorithms for critical-care enteral and parenteral therapy (ACCEPT). CMAJ. 2004 Jan 20;170(2):197-204. PMID 14734433
- [Background] Jain MK, Heyland D, Dhaliwal R, Day AG, Drover J, Keefe L, Gelula M. Dissemination of the Canadian clinical practice guidelines for nutrition support: results of a cluster randomized controlled trial. Crit Care Med. 2006 Sep;34(9):2362-9. doi: 10.1097/01.CCM.0000234044.91893.9C. PMID 16850001
- [Background] Heyland DK, Murch L, Cahill N, McCall M, Muscedere J, Stelfox HT, Bray T, Tanguay T, Jiang X, Day AG. Enhanced protein-energy provision via the enteral route feeding protocol in critically ill patients: results of a cluster randomized trial. Crit Care Med. 2013 Dec;41(12):2743-53. doi: 10.1097/CCM.0b013e31829efef5. PMID 23982032
- [Background] Cahill NE, Dhaliwal R, Day AG, Jiang X, Heyland DK. Nutrition therapy in the critical care setting: what is "best achievable" practice? An international multicenter observational study. Crit Care Med. 2010 Feb;38(2):395-401. doi: 10.1097/CCM.0b013e3181c0263d. PMID 19851094
- [Background] Heyland DK, Dhaliwal R, Wang M, Day AG. The prevalence of iatrogenic underfeeding in the nutritionally 'at-risk' critically ill patient: Results of an international, multicenter, prospective study. Clin Nutr. 2015 Aug;34(4):659-66. doi: 10.1016/j.clnu.2014.07.008. Epub 2014 Jul 19. PMID 25086472
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Ferguson M, Capra S, Bauer J, Banks M. Development of a valid and reliable malnutrition screening tool for adult acute hospital patients. Nutrition. 1999 Jun;15(6):458-64. doi: 10.1016/s0899-9007(99)00084-2. PMID 10378201
- [Background] Baker JP, Detsky AS, Wesson DE, Wolman SL, Stewart S, Whitewell J, Langer B, Jeejeebhoy KN. Nutritional assessment: a comparison of clinical judgement and objective measurements. N Engl J Med. 1982 Apr 22;306(16):969-72. doi: 10.1056/NEJM198204223061606. No abstract available. PMID 6801515
- [Background] Faisy C, Lerolle N, Dachraoui F, Savard JF, Abboud I, Tadie JM, Fagon JY. Impact of energy deficit calculated by a predictive method on outcome in medical patients requiring prolonged acute mechanical ventilation. Br J Nutr. 2009 Apr;101(7):1079-87. doi: 10.1017/S0007114508055669. Epub 2008 Sep 9. PMID 18778528
- [Background] Moisey LL, Mourtzakis M, Cotton BA, Premji T, Heyland DK, Wade CE, Bulger E, Kozar RA; Nutrition and Rehabilitation Investigators Consortium (NUTRIC). Skeletal muscle predicts ventilator-free days, ICU-free days, and mortality in elderly ICU patients. Crit Care. 2013 Sep 19;17(5):R206. doi: 10.1186/cc12901. PMID 24050662
- [Background] Malmstrom TK, Morley JE. SARC-F: a simple questionnaire to rapidly diagnose sarcopenia. J Am Med Dir Assoc. 2013 Aug;14(8):531-2. doi: 10.1016/j.jamda.2013.05.018. Epub 2013 Jun 25. No abstract available. PMID 23810110
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Background] Committee for Proprietary Medicinal Products (CPMP). Committee for Proprietary Medicinal Products (CPMP): points to consider on adjustment for baseline covariates. Stat Med. 2004 Mar 15;23(5):701-9. doi: 10.1002/sim.1647. No abstract available. PMID 14981670
- [Background] International conference on harmonisation; guidance on statistical principles for clinical trials; availability--FDA. Notice. Fed Regist. 1998 Sep 16;63(179):49583-98. PMID 10185190
- [Background] Kahan BC. Accounting for centre-effects in multicentre trials with a binary outcome - when, why, and how? BMC Med Res Methodol. 2014 Feb 10;14:20. doi: 10.1186/1471-2288-14-20. PMID 24512175
- [Background] Gray RJ. A class of $ K $-sample tests for comparing the cumulative incidence of a competing risk. The Annals of statistics 1988;16(3):1141-54.
- [Background] Duchateau L, Janssen P, Lindsey P, et al. The shared frailty model and the power for heterogeneity tests in multicenter trials. Computational Statistics & Data Analysis 2002;40(3):603-20.
- [Background] Liublinska V, Rubin DB. Sensitivity analysis for a partially missing binary outcome in a two-arm randomized clinical trial. Stat Med. 2014 Oct 30;33(24):4170-85. doi: 10.1002/sim.6197. Epub 2014 May 20. PMID 24845086
- [Background] Hollis S. A graphical sensitivity analysis for clinical trials with non-ignorable missing binary outcome. Stat Med. 2002 Dec 30;21(24):3823-34. doi: 10.1002/sim.1276. PMID 12483769
- [Background] Gordon Lan K, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika 1983;70(3):659-63.
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Fine JP, Gray RJ. A proportional hazards model for the subdistribution of a competing risk. Journal of the American statistical association 1999;94(446):496-509.
- [Background] Faden RR, Kass NE, Goodman SN, Pronovost P, Tunis S, Beauchamp TL. An ethics framework for a learning health care system: a departure from traditional research ethics and clinical ethics. Hastings Cent Rep. 2013 Jan-Feb;Spec No:S16-27. doi: 10.1002/hast.134. No abstract available. PMID 23315888
- [Background] Faden RR, Beauchamp TL, Kass NE. Informed consent, comparative effectiveness, and learning health care. N Engl J Med. 2014 Feb 20;370(8):766-8. doi: 10.1056/NEJMhle1313674. No abstract available. PMID 24552325
- [Background] Truog RD, Robinson W, Randolph A, Morris A. Is informed consent always necessary for randomized, controlled trials? N Engl J Med. 1999 Mar 11;340(10):804-7. doi: 10.1056/NEJM199903113401013. No abstract available. PMID 10072420
- [Background] Faden R, Kass N, Whicher D, Stewart W, Tunis S. Ethics and informed consent for comparative effectiveness research with prospective electronic clinical data. Med Care. 2013 Aug;51(8 Suppl 3):S53-7. doi: 10.1097/MLR.0b013e31829b1e4b. PMID 23793051
- [Background] Kim SY, Miller FG. Informed consent for pragmatic trials--the integrated consent model. N Engl J Med. 2014 Feb 20;370(8):769-72. doi: 10.1056/NEJMhle1312508. No abstract available. PMID 24552326
- [Background] Semler MW, Wanderer JP, Ehrenfeld JM, Stollings JL, Self WH, Siew ED, Wang L, Byrne DW, Shaw AD, Bernard GR, Rice TW; SALT Investigators * and the Pragmatic Critical Care Research Group; SALT Investigators. Balanced Crystalloids versus Saline in the Intensive Care Unit. The SALT Randomized Trial. Am J Respir Crit Care Med. 2017 May 15;195(10):1362-1372. doi: 10.1164/rccm.201607-1345OC. PMID 27749094
- [Background] Janz DR, Semler MW, Lentz RJ, Matthews DT, Assad TR, Norman BC, Keriwala RD, Ferrell BA, Noto MJ, Shaver CM, Richmond BW, Zinggeler Berg J, Rice TW; Facilitating EndotracheaL intubation by Laryngoscopy technique and apneic Oxygenation Within the ICU Investigators and the Pragmatic Critical Care Research Group. Randomized Trial of Video Laryngoscopy for Endotracheal Intubation of Critically Ill Adults. Crit Care Med. 2016 Nov;44(11):1980-1987. doi: 10.1097/CCM.0000000000001841. PMID 27355526
- [Background] Semler MW, Janz DR, Lentz RJ, Matthews DT, Norman BC, Assad TR, Keriwala RD, Ferrell BA, Noto MJ, McKown AC, Kocurek EG, Warren MA, Huerta LE, Rice TW; FELLOW Investigators; Pragmatic Critical Care Research Group. Randomized Trial of Apneic Oxygenation during Endotracheal Intubation of the Critically Ill. Am J Respir Crit Care Med. 2016 Feb 1;193(3):273-80. doi: 10.1164/rccm.201507-1294OC. PMID 26426458
- [Background] Canadian Critical Care Trials Group. A randomized trial of diagnostic techniques for ventilator-associated pneumonia. N Engl J Med. 2006 Dec 21;355(25):2619-30. doi: 10.1056/NEJMoa052904. PMID 17182987
- [Background] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003